CLINICAL TRIAL: NCT03834558
Title: SarcoImage: Anatomical and Physiological Validation by Magnetic Resonance Imaging Biomarkers of the Effects of High Intensity Strenght Training and Myofascial Self-conditioning on Sarcopenia in Frail and Prefrail Elderly
Brief Title: Imaging Biomarkers of the Effects of a Mixed Exercise Program
Acronym: SarcoImage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Fundación Universidad Católica de Valencia San Vicente Mártir (Other); Quironsalud (Other)
Responsible Party: Principal Investigator, Francisco Martínez Arnau, Martínez-Arnau FM, PT, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1488746567568
Record Dates: First submitted 2018-09-24; First posted 2019-02-08 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Frailty; Strength; myofascial self conditioning; image biomarkers
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Intervention Model Description: This project is based on an, longitudinal, prospective, controlled, randomized, intervention study and blind for the researchers responsible for the study. Thus, the subjects participating in the study will be divided into 2 groups, one of which will perform the mixed exercise program (intervention group, IG), and another that will follow their daily routine without added exercise (control group, CG).
  Each group will have 2 measurements in which the corresponding variables will be evaluated: A) before the start of the intervention, B) at 6 months (at the end of the intervention)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator: The persons who make the data analysis and decide whether a patient has experienced an outcome of interest will be masked.
  Outcome assessors: The persons who assess patients and provide outcome data will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): They will follow their daily routine without added exercise
- Intervention Group (Experimental): They will perform the mixed exercise program
  Interventions: Other: Mixed exercise program

INTERVENTIONS:
Other: Mixed exercise program — A progressive program of high intensity strength and myofascial conditioning will be carried out in 2 non-consecutive weekly sessions (24 weeks). Each session will include:
  A) Warm up on a cycle ergometer
  B) Strength circuit: 6 exercises will be included to strengthen different muscle groups (2 in the upper extremities, 2 in the trunk and 2 in the lower extremities). 3 sets of 10-15 repetitions until the failure. The load will be set to 70% of 1 maximal resistance.
  C) Self-myofascial conditioning: 10 repetitions, in the direction of the fibres of each muscle group, with different materials. 7 muscle groups will be worked (quadriceps, hamstrings, abductors, gluteus, pectoralis, full back and trapezius).
  D) At the end, static stretches will be performed
  Arms: Intervention Group

SUMMARY:
The aim is quantify, correlate and establish the diagnostic and prognostic value of the variation of the image biomarkers obtained by magnetic resonance (muscle volume, morphological, biochemical and structural biomarkers) longitudinally in fragile or pre-frail elders with sarcopenia after a mixed physical training of strength and myofascial self-conditioning. This project is based on an, longitudinal, prospective, controlled, randomized, intervention study and blind for the researchers responsible for the study. 60 elderly with sarcopenia and frailty (Intervention Group, n=30; Control Group, n=30) will participate in the study. Intervention Group participants will perform 6-months mixed exercise program consisting in high-intensity strength training and self-myofascial conditioning. Data will be take trough 2 measurements that will be take place at baseline and post-intervention. Criteria of frailty, criteria of sarcopenia, sociodemographic, clinics, kinanthropometric, functional, nutritional and confusing variables will be evaluated. Moreover, magnetic resonance images will be performed to obtain muscle volume, morphological, biochemical and structural biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders,
* aged 70 years old or more,
* with habitual residence in Valencia,
* with independent wandering (they can have technical aids, but not from someone else)
* that meets Fried's pre-frailty or frailty criteria
* EGWSOP's sarcopenia criteria
* who has agreed to participate in the study and signed the informed consent

Exclusion Criteria:

* Patients with life expectancy less than six months
* Institutionalized patients
* Patients with severe visual or auditory deficits
* Patients with contraindication in the performance of physical exercise (cardiovascular risk factors)
* Patients with contraindications for the magnetic resonance study, especially carriers of non-compatible pacemakers, neurostimulators, cochlear implants and intracranial aneurysm clamping.
* Patients with severe psychiatric illness or moderate or severe cognitive impairment.
* Patients who refuse to sign the informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Muscle volume | 6 months
  Changes related to macroscopic changes in muscle tissue assessed by magnetic resonance after a 6-month program of high intensity training and myofascial self-conditioning, specifically muscle volume of the thigh by compartment - anterior, medial and posterior (in ml)
Bone volume | 6 months
  Changes related to macroscopic changes in bone tissue assessed by magnetic resonance after a 6-month program of high intensity training and myofascial self-conditioning, specifically relative volume of bone (in %)
Relative volume of intramuscular fat | 6 months
  Changes related to macroscopic changes in fat tissue assessed by magnetic resonance after a 6-month program of high intensity training and myofascial self-conditioning, specifically relative volume of intramuscular fat (in %)
Extramuscular subcutaneous fat | 6 months
  Changes related to macroscopic changes in fat tissue assessed by magnetic resonance after a 6-month program of high intensity training and myofascial self-conditioning, specifically extramuscular subcutaneous fat (in ml)
Microscopic fat fraction | 6 months
  Changes related to microscopic changes in fat tissue assessed by magnetic resonance after a 6-month program of high intensity training and myofascial self-conditioning, specifically microscopic fat fraction (in %)
Descriptors of muscle texture | 6 months
  Changes related to microscopic changes in muscle tissue assessed by magnetic resonance after a 6-month program of high intensity training and myofascial self-conditioning, specifically statistical descriptors of muscle texture: energy, entropy, contrast and homogeneity (adimensional)
Diffusion coefficient | 6 months
  Changes related to microscopic changes in diffusion coefficient assessed by magnetic resonance after a 6-month program of high intensity training and myofascial self-conditioning, specifically diffusion coefficient and apparent diffusion coefficient (mm2/s)

SECONDARY OUTCOMES:
Body muscle mass | 6 months
  Changes produced by 6-month program of high intensity training and myofascial self-conditioning on body muscle mass (kg/m2) measured according to criteria of sarcopenia of European Working Group of Sarcopenia in Older People.
Handgrip strength | 6 months
  Changes produced by 6-month program of high intensity training and myofascial self-conditioning on handgrip strength (kg) measured according to criteria of sarcopenia of European Working Group of Sarcopenia in Older People.
Walking speed | 6 months
  Changes produced by 6-month program of high intensity training and myofascial self-conditioning on walking speed (m/s) measured according to criteria of sarcopenia of European Working Group of Sarcopenia in Older People.
Body mass index | 6 months
  Changes on body mass index (measured in kg/m2) generated by 6-month program of high intensity training and myofascial self-conditioning
Lean mass | 6 months
  Changes on lean impedance (measured in % by bioimpedance) generated by 6-month program of high intensity training and myofascial self-conditioning
Fat mass | 6 months
  Changes on fat impedance (measured in % by bioimpedance) generated by 6-month program of high intensity training and myofascial self-conditioning
Body perimeters | 6 months
  Changes on calf and thigh perimeter (measured in cm) generated by 6-month program of high intensity training and myofascial self-conditioning
Articular range | 6 months
  Changes on range of joint movement of coxofemoral and knee articulation (measured in degrees) generated by 6-month program of high intensity training and myofascial self-conditioning
Perceived pain | 6 months
  Changes on pain (measured by visual analogic scale, 0 to 10 points, higher values = worse outcome) generated by 6-month program of high intensity training and myofascial self-conditioning
Activities of daily living | 6 months
  Changes in functionality and independence measured by Barthel Index (0 to 100 points, < 60 dependence, higher values = better outcome) produced by 6-month program of high intensity training and myofascial self-conditioning
Functional and physical performance | 6 months
  Changes in functional and physical performance measured by Short Physical Performance Battery (0 to 12 points, higher score = higher function) produced by 6-month program of high intensity training and myofascial self-conditioning
Forced spirometry | 6 months
  Changes in respiratory function, measured by forced spirometry parameters assessed with a spirometer, produced by 6-month program of high intensity training and myofascial self-conditioning
Respiratory muscles strength | 6 months
  Changes in respiratory pressures generated in mouth by respiratory muscles (assessed with a respiratory pressure gauge) produced by 6-month program of high intensity training and myofascial self-conditioning
Perceived quality of life | 6 months
  Changes produced by 6-month program of high intensity training and myofascial self-conditioning related to quality of life (EuroQol 5 Dimensions - 3 levels Index, 0 to 1 points, higher values = better outcome)
Type of drugs used | 6 months
  Type and dose of drugs consumed before and after a 6-month program of high intensity training and myofascial self-conditioning

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Martinez Arnau, PhD, Principal Investigator — Universitat de Valencia; Roberto Sanz Requena, PhD, Study Director — Hospital QuironSalud - Hospital Universitario La Fe (GIBI); Ana Pablos Monzó, PhD, Study Director — Fundación Universidad Católica de Valencia; Pilar Pérez-Ros, PhD, Study Director — Fundación Universidad Católica de Valencia
Locations (1):
- University of Valencia - Faculty of Physiotherapy, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers

REFERENCES:
- [Derived] Flor-Rufino C, Barrachina-Igual J, Perez-Ros P, Pablos-Monzo A, Sanz-Requena R, Martinez-Arnau FM. Fat infiltration and muscle hydration improve after high-intensity resistance training in women with sarcopenia. A randomized clinical trial. Maturitas. 2023 Feb;168:29-36. doi: 10.1016/j.maturitas.2022.09.001. Epub 2022 Nov 4. PMID 36423489
- [Derived] Flor-Rufino C, Barrachina-Igual J, Perez-Ros P, Pablos-Monzo A, Martinez-Arnau FM. Resistance training of peripheral muscles benefits respiratory parameters in older women with sarcopenia: Randomized controlled trial. Arch Gerontol Geriatr. 2023 Jan;104:104799. doi: 10.1016/j.archger.2022.104799. Epub 2022 Aug 29. PMID 36070636